CLINICAL TRIAL: NCT03750032
Title: Technical Modifications of Appendicular Stump Closure During Laparoscopic Appendectomy
Acronym: CAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-CHIR-CAS
Record Dates: First submitted 2018-11-02; First posted 2018-11-21 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Acute Appendicitis
Keywords: acute appendicitis; laparoscopy; closure of appendicular stump; economical and medical outcomes
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Intervention Model Description: The patients will be randomized into three groups of various appendicular stump closure.
Masking Description: No masking will be used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stapler appendectomy (Experimental): A total of 40 study subjects undergoing appendectomy will be randomized into the group with appendicular stump closure using a stapler.
  Interventions: Procedure: Stapler appendectomy
- Endoloop (Experimental): A total of 40 study subjects undergoing appendectomy will be randomized into the group with appendicular stump closure using endoloop.
  Interventions: Procedure: Endoloop
- Hem-O-Lock (Experimental): A total of 40 study subjects undergoing appendectomy will be randomized into the group with appendicular stump closure using Hem-O-Lock.
  Interventions: Procedure: Hem-O-Lock

INTERVENTIONS:
Procedure: Stapler appendectomy — The patients randomised for this intervention will undergo stapler appendectomy.
  Arms: Stapler appendectomy
Procedure: Endoloop — The patients randomised for this intervention will undergo appendicular stump closure using Endoloop.
  Arms: Endoloop
Procedure: Hem-O-Lock — The patients randomised for this intervention will undergo appendicular stump closure using Hem-O-Lock.
  Arms: Hem-O-Lock

SUMMARY:
Laparoscopic appendectomy (L-APPE) presents a golden standard in the treatment of acute appendicitis nowadays. However, there are ongoing controversies regarding the ideal technique of appendicular stump closure during L-APPE in the published literature. Several technical modifications of appendicular stump closure are available at the present - closure using endoloop, endostapler or Hem-o-lock clips. The aim of the proposed project (CAS study) is to compare medical and economic outcomes of patients undergoing L-APPE with different methods of appendicular stump closure (endostapler, endoloop and Hem-o-lock clips).

DETAILED DESCRIPTION:
Acute appendicitis presents one of the most common surgical illnesses which affect approximately 7% of the western population. In the Czech Republic, 11664 patients were hospitalized and operated for the diagnosis of acute appendicitis (K35-K38) during 2016. It might seem that the procedure of appendectomy will be guided by a clear algorithm for its frequency, but it is not so. Because of acute appendicitis, appendectomy may be performed via laparotomy or laparoscopy (minimally invasive surgery). During laparoscopic appendectomy (L-APPE), there are no clear recommendations regarding trocar placement, methods of dividing appendicular mesenteriolum, methods of appendicular stump closure or appendicular stump sinking.

The proposed clinical study is focused on the issue of the appendicular base interruption during L-APPE. At the present, there are several technical modifications of appendicular stump closure - by means of endoloop (the suture loop from absorbable fiber), endostapler or using Hem-o-lock clips. The performed literature search revealed that evidence-based medicine data regarding the optimal way of appendicular stump closure are insufficient. That is why the investigators have decided to conduct a prospective randomized single-center clinical study aimed to compare different technical modifications of appendicular stump closure during L-APPE. Within a study period, all patients undergoing L-APPE at the University Hospital Ostrava will be randomized to one of the technical modifications of appendicular stump closure.

The aim of the project (CAS study) is to compare medical and economic outcomes of patients undergoing L-APPE with different methods of appendicular stump closure (endostapler, endoloop and Hem-o-lock clips). The operative time, intraoperative and postoperative complications will be the primary outcome measures of the study, economic outcomes will be the secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* acute appendicitis
* laparoscopic approach
* signed informed content

Exclusion Criteria:

- necrosis or advanced inflammatory changes in the area of appendicular stump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Operative time | 12 months
  Operative time will be measured in minutes and analysed.
Incidence of intraoperative and postoperative complications | 12 months
  The incidence of intraoperative and postoperative complications will be analysed in all groups of study subjects.

SECONDARY OUTCOMES:
Costs of surgery | 12 months
  Costs of surgery will be analysed for all groups of study subjects.
Costs of hospitalization | 12 months
  The overall costs of hospitalisation will be analysed for all groups of study subjects.
Costs of treatment of complications | 12 months
  Costs of treatment of complications will be analysed for all groups of study subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ihnát, Ass.Prof.,MD,PhD,MBA, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not decided to make the individual participant data available to other researchers.

REFERENCES:
- [Background] Mayir B, Bilecik T, Ensari CO, Oruc MT. Laparoscopic appendectomy with hand-made loop. Wideochir Inne Tech Maloinwazyjne. 2014 Jun;9(2):152-6. doi: 10.5114/wiitm.2014.41624. Epub 2014 Mar 24. PMID 25097680
- [Background] Matyja M, Strzalka M, Rembiasz K. Laparosocopic Appendectomy, Cost-Effectiveness of Three Different Techniques Used to Close the Appendix Stump. Pol Przegl Chir. 2015 Dec;87(12):634-7. doi: 10.1515/pjs-2016-0015. PMID 26963058
- [Background] Mayir B, Ensari CO, Bilecik T, Aslaner A, Oruc MT. Methods for closure of appendix stump during laparoscopic appendectomy procedure. Ulus Cerrahi Derg. 2015 Aug 18;31(4):229-31. doi: 10.5152/UCD.2015.2768. eCollection 2015. PMID 26668532
- [Background] Yildiz I, Koca S. Is There An Ideal Stump Closure Technique In Laparoscopic Appendectomy? Surg Technol Int. 2016 Apr;28:117-20. PMID 27121413
- [Background] Delibegovic S, Mehmedovic Z. Erratum to: The Influence of the Appendiceal Base Diameter on Appendix Stump Closure in Laparoscopic Appendectomy. World J Surg. 2016 Nov;40(11):2832. doi: 10.1007/s00268-016-3709-5. No abstract available. PMID 27627887
- [Derived] Ihnat P, Tesar M, Tulinsky L, Ihnat Rudinska L, Okantey O, Durdik S. A randomized clinical trial of technical modifications of appendix stump closure during laparoscopic appendectomy for uncomplicated acute appendicitis. BMC Surg. 2021 May 31;21(1):272. doi: 10.1186/s12893-021-01279-z. PMID 34059039